CLINICAL TRIAL: NCT03084263
Title: A Comparison Study of Arthroscopic Assisted Open Reduction Internal Fixation (AORIF) Versus Open Reduction Internal Fixation (ORIF) in Ankle Fractures: Does AORIF Improve Functional Outcomes?
Brief Title: Arthroscopic Assisted Open Reduction Internal Fixation Versus Open Reduction Internal Fixation in Ankle Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn (No Participants Enrolled)
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-061
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AORIF of Ankle Fractures (Experimental): Arthroscopic Assisted Open Reduction Internal Fixation of ankle fracture.
  Interventions: Procedure: Arthroscopic Assisted Open Reduction Internal Fixation
- ORIF of Ankle Fractures (Active Comparator): Open Reduction Internal Fixation of ankle fracture.
  Interventions: Procedure: Open Reduction Internal Fixation

INTERVENTIONS:
Procedure: Arthroscopic Assisted Open Reduction Internal Fixation — Surgical fixation of ankle fractures with use of arthroscopy.
  Other Names: AORIF
  Arms: AORIF of Ankle Fractures
Procedure: Open Reduction Internal Fixation — Surgical fixation of ankle fractures.
  Other Names: ORIF
  Arms: ORIF of Ankle Fractures

SUMMARY:
The objective of this study is to compare the functional outcomes of patients with ankle fractures treated by Arthroscopic assisted Open Reduction Internal Fixation (AORIF) versus Open Reduction Internal Fixation (ORIF).

DETAILED DESCRIPTION:
Prospective Randomized Clinical Trial evaluating patients with ankle fractures undergoing AORIF versus ORIF

Participants will be randomized into 2 different surgical groups, one group receiving only ORIF and the other group receiving AORIF.

As standard of care patients will follow up in the office at approximately 3 weeks, 6 weeks and 12 weeks post operatively. Patients will be immobilized in a splint and will be non-weight bearing until their 3 week post-op visit. At the 3 week post-op visit, the patient will be fitted in a boot, be instructed to begin self-directed ROM and to continue non-weight bearing. At the 6 week post-op visit, the patient will begin weight bearing in the boot.

In office study visit will occur at these same times. At each visit weight bearing status, return to sports, pain level, AOFAS and FAAM will be assessed. One additional study visit will be conducted over the phone or by mail at approximately one year post operatively and will consist of the FAAM.

ELIGIBILITY:
Inclusion Criteria:

* Closed ankle fractures (44A, 44B, 44C)
* Ages of 18-65
* Men or women, including pregnant women
* Willing to consent

Exclusion Criteria:

* Open fractures
* Other lower extremity injuries/conditions that affects functional outcomes
* Problems maintaining follow up (homeless, not willing to return for follow up)
* Prisoners
* Unable to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Score (AOFAS) | 6 month
  Compare AOFAS scores between AORIF versus ORIF of ankle fractures.
Foot and Ankle Ability Measure (FAAM) | 1 year
  Compare FAAM scores between AORIF versus ORIF of ankle fractures.
Rate of Return to Sports | 1 year
  Compare Return to Sports rates between AORIF versus ORIF of ankle fractures.

SECONDARY OUTCOMES:
Rates of Complications | 1 year
  Compare rates of Complication between AORIF versus ORIF of ankle fractures.
Pain Scores | 1 year
  Compare Pain Scores between AORIF versus ORIF of ankle fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Anderson, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No